CLINICAL TRIAL: NCT06575829
Title: Open Label, Single-center Pilot Study to Investigate Alglucosidase Alfa (20 mg/kg) Frequency Reduction From 2 to 4 Weeks in a Subgroup of Elderly Patients With Late-onset Pompe Disease (TRIPOD-Study)
Brief Title: Treatment Frequency Reduction in Pompe Disease
Acronym: TRIPOD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ina Barzel, Coordinating investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL99999.999.99; 2024-514255-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pompe Disease (Late-onset); GAA Deficiency; Glycogen Storage Disease Type II; Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Intervention Model Description: This study is a self-controlled cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Algucosidase alfa 20 mg/kg once every 4 weeks instead of once every 2 weeks (Experimental): Alglucosidase alfa will be administered by intravenous infusion at a dose of 20 mg/kg once every 4 weeks instead of once every 2 weeks for a duration of 9 months.
  After 9 months of treatment with the extended interval, it will be determined for each patient whether it is considered safe to discontinue enzyme replacement therapy (ERT). Both, patients who stop ERT after 9 months and those who continue with either the new or the previous dosing schedule, will be closely followed for an additional 12 months, leading to a total study duration of 21 months.
  Interventions: Drug: Algucosidase alfa 20 mg/kg once every 4 weeks instead of once every 2 weeks

INTERVENTIONS:
Drug: Algucosidase alfa 20 mg/kg once every 4 weeks instead of once every 2 weeks — The interval of ERT with alglucosidase alfa will be extended from once every 2 weeks to once every 4 weeks. The dose of 20 mg/kg per infusion remains the same.

SUMMARY:
The aim of this study is to assess if dosing frequency reduction of alglucosidase alfa 20 mg/kg once every 2 weeks to once every 4 weeks is safe and does not lead to increased progression of disease in a selected group of patients with late-onset Pompe disease.

DETAILED DESCRIPTION:
All eligible patients with late-onset Pompe disease will be treated with alglucosidase alfa 20 mg/kg once every 4 weeks for 9 months. During the study, patients will be monitored once every 3 months.

After 9 months of treatment with the extended interval, it will be determined for each patient whether it is considered safe to discontinue enzyme replacement therapy (ERT). The investigators consider it safe: 1] if the patient is stable compared to the year prior to reducing the ERT frequency, or, 2] if the patient previously deteriorated (slightly) despite standard ERT and this deterioration is not exaggerated by the alternative dosing regimen. If after 9 months there is no valid medical reason to switch back to standard dosing (once every 2 weeks) and the patient does not wish to discontinue treatment, the 4-week dosing regimen will be continued. If at any moment a patient shows an unexpectedly rapid decline in clinical outcome parameters (significantly higher than their own course at regular treatment dosage), treatment will be switched back to or be restarted with the standard dosing regimen of 20 mg/kg every 2 weeks.

Both, patients who stop ERT after 9 months and those who continue with either the new or the previous dosing schedule, will be closely followed for an additional 12 months to be able to take action (e.g., switch to a standard dosing regimen or restart ERT) if a more rapid clinical deterioration occurs than expected, or to investigate if muscle and pulmonary function regain when standard dosage has been re-instituted after signs of clinical deterioration during the 4-week treatment interval. After the end of the study (21 months), patients will be carefully followed according to the standard frequency (once every 6 months). If a patient shows an unexpectedly rapid decline in clinical outcome parameters henceforth, treatment will be switched back to or be restarted with the standard dosing regimen of 20 mg/kg eow.

ELIGIBILITY:
Inclusion Criteria:

* LOPD (confirmed diagnosis: enzyme deficiency in any tissue source and/or 2 confirmed disease-causing variants in the GAA gene)
* Age ≥50 years
* Current treatment with alglucosidase alfa at a standard dose of 20 mg/kg once every 2 weeks for ≥4 years
* Relatively stable clinical condition over the past year
* Able to walk ≥150 m within 6 minutes (6MWT)
* (Forced) vital capacity (FVC) in sitting position: >55% of expected value and in supine position: >45% of expected value
* Willing and able to adhere to the study procedures

Exclusion Criteria:

* Rapidly progressive muscle weakness
* Severely limited muscle strength almost requiring/requiring daily wheelchair use
* Requiring respiratory support (non-invasive/invasive ventilation) or being at high risk to require respiratory support (ventilation) due to further deterioration of current pulmonary function. Using continuous positive airway pressure (CPAP) support only for obstructive sleep apnea syndrome (OSAS) is permitted.
* Comorbidities which are expected to influence the primary outcome measures within the next 2 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle strength and function by manual muscle testing with Medical Research Council (MRC) grading scale | At baseline and every 3 months for a duration of 21 months.
  Muscle strength will be determined by manual muscle testing using the Medical Research Council (MRC) grading scale. Muscle strength is graded from 0-5 by physical examination, in which grade 5 represents normal muscle strength and grade 0 means paralysis of the muscle group tested. Muscle groups tests will include neck flexors/extensors, shoulder abductors, elbow extensors/flexors, wrist extensors/flexors, hip extension, hip flexors, hip adductors/abductors, knee extensors/flexors, and foot extensors/flexors.
Changes in muscle strength and function by testing hand-held dynamometry (HHD) | At baseline and every 3 months for a duration of 21 months.
  Muscle strength will be measured with the CITEC hand-held dynamometer (HHD). Thirteen muscle groups will be tested: neck extension, neck flexion, and bilateral shoulder abduction, elbow flexion, elbow extension, wrist extension, squeezing, hip flexion, hip extension, hip abduction, knee flexion, knee extension, ankle dorsiflexion, and ankle plantar flexion. A mean value in Newton (N) is calculated from three consecutive measurements per muscle group.
Changes in muscle strength and function by quick motor function test (QMFT) | At baseline and every 3 months for a duration of 21 months.
  The QMFT will be administered at the time points specified. This 16-item functional test has been developed to evaluate the function of the muscle groups that are specifically affected in patients with Pompe disease. The patient is asked to perform multiple activities in supine, sitting and standing position. The performance of the patient is scored on a 5-point ordinal scale (range 0-4). This standardized test can be performed within 5-10 minutes and can be performed in children and adults with varying disease severity.
Changes in muscle strength and function by 6-minute walk test (6MWT) | Every 3 months for a duration of 21 months.
  The 6MWT is a timed test that measures functional endurance. The primary measurement is the distance walked in 6 minutes, measured in meters. The percent of predicted distance and the amount of time walked (to quantify endurance, as not all patients may complete the full 6-minute walk) will also be recorded. The patient is instructed to walk the length of a pre-measured hallway for six minutes. It is widely regarded as an objective measure, which is easy to perform and reflects the performance in ADL of the patient.
Changes in pulmonary function by testing forced vital capacity (FVC) in sitting and supine positions | At baseline and every 3 months for a duration of 21 months.
  Pulmonary function testing will be performed at the time points specified. Forced vital capacity will be measured during sitting and supine positions as a measure of lung volume (and indirect measure of the strength of the diaphragm and abdominal muscles).
  The pulmonary testing protocol is standardized in accordance with ATS/ERS Guidelines36.
  Three repeated reproducible flow volume curves will be made. The best effort will be used for further analyses. Values will be expressed as a percentage of the predicted normal values or as z-score, based on age, gender, race, and height. Global Lung Initiative (GLI) 2012 reference equations will be used.
Changes in pulmonary function by testing maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) | At baseline and every 3 months for a duration of 21 months.
  In addition to the vital capacity, inspiratory (MIP) and expiratory (MEP) mouth pressures will be measured in upright seated position to determine the maximum force that can be exerted by the respiratory muscles.
  MIP will be measured at residual volume after maximal expiration, while MEP is registered at total lung capacity after maximal inspiration. Pressures must be maintained at least 1 second. Maneuvers will be repeated until three reproducible methods are obtained. The highest value will be taken for analyses.
Changes in patient reported outcome measures by filling in the Rasch-built Pompe-specific activity (R-PAct) scale | At baseline and every 3 months for a duration of 21 months.
  The Rasch-built Pompe-specific activity (R-PAct) scale is a self-reported, 18-items questionnaire designed specifically for use in patients with Pompe disease, based upon experiences from patients about their most important and limiting aspects in daily life. All items have three response options: [0] unable to perform; [1] able to perform, but with difficulty or [2] able to perform without difficulty. If all items are answered, an appropriate centile metric score (range 0-100) will be calculated.
Changes in patient reported outcome measures by filling in the SF-36 questionnaire | At baseline, after 9 months and at the end of the study (21 months).
  The SF-36 is a health-related quality of life questionnaire, consisting of 36 items. The items are assigned to the domains of physical functioning, role functioning-physical, role functioning-emotional, social functioning, body pain, mental health, vitality, general health perception and change in health.
Body weight | At baseline and every 3 months for a duration of 21 months.
  Body weight will be measured in kilograms (kg).
Heart rate | At baseline and every 4 weeks at the start and at the end of the aglucosidase alfa infusion for a duration of 9 months. If alglucosidase alfa treatment is not stopped after 9 months, the measurement will take place for a total duration of 21 months.
  Heart rate will be measured in beats per minute (bpm).
Systolic and diastolic blood pressure | At baseline and every 4 weeks at the start and at the end of the aglucosidase alfa infusion for a duration of 9 months. If alglucosidase alfa treatment is not stopped after 9 months, the measurement will take place for a total duration of 21 months.
  Systolic and diastolic blood pressure will be measured in millimeter of mercury (mmHg).
Respiratory rate | At baseline and every 4 weeks at the start of the aglucosidase alfa infusion for a duration of 9 months. If alglucosidase alfa treatment is not stopped after 9 months, the measurement will take place for a total duration of 21 months.
  Respiratory rate will be measured in breaths per minute.

SECONDARY OUTCOMES:
Changes in lean body mass assessed by DEXA-scans | At baseline, after 9 months and at the end of the study (21 months).
  Body composition will be measured conform DEXA technology (currently at Erasmus MC: GE Healthcare Lunar iDXA equipment: densitometer and encore software). This is a low-cost technology and simultaneously accurate, easy to perform and involves very low radiation dose (8 µSv per scan) to the patient which brings no harm. This imaging technique is the gold standard technique for the assessment of body composition.
  Body composition will be presented as mineral bone, fat and fatty free body mass in kilograms.
Changes in lean body mass assessed by DEXA-scans | At baseline, after 9 months and at the end of the study (21 months).
  Percentages of total body fat mass, android and gynoid fat will be measured. Percentages of fat mass will also be measured at regional level (arms, trunk and legs).
Bone density assessed by DEXA-scans | At baseline, after 9 months and at the end of the study (21 months).
  Bone mineral density is measured at total body in g/cm2.
Need for walking devices and artificial ventilation (yes/no) | At baseline and every 3 months for a duration of 21 months.
  For the purpose of stabilization and if deemed necessary by the investigator, the patient may use a walking device during the assessment, such as cane or walker. If such a device is used during the assessment, this must be recorded in the CRF/HiX. It will also be determined whether patients may need non-invasive or invasive ventilation during the study, including the hours of ventilation per day.
Changes in alglucosidase alfa activity in plasma | At 3 months and 9 months.
  Blood samples will be collected before and after infusion of alglucosidase alfa at week 13 and week 39. Sampling times are as follows: pre-dose, 15 minutes before end of infusion, directly after end of infusion and 9 hours after start of infusion. The activity of alglucosidase alfa will be analyzed by the clinical chemistry laboratory of the Erasmus MC and expressed as nanomol 4-methylumbelliferyl-α-glucopyranoside (MU)/hour/10 microliter.
Serological testing of serum creatine kinase (CK) and antibodies against alglucosidase alfa | At baseline and every 3 months for a duration of 21 months.
  Blood samples will be drawn at baseline and at every 3 months for determination of serum creatine kinase (CK). Potential antibodies against alglucosidase alfa will be determined at baseline, after 9 months and at the end of the study (21 months).
Urine tetraglucoside | At baseline and every 3 months for a duration of 21 months.
  Urine tetraglucoside (Glc4) will be measured in micromol/millimol kreatinine.
Assessment of treatment-emergent adverse events (TEAEs), including infusion associated reactions (IARs) | At baseline and every 3 months for a duration of 21 months.
  At each study visit, patients will be evaluated for new TEAEs in regard to the intervention (extension of the dosing interval, possibly followed by discontinuation of therapy). Adverse events potentially associated with (accelerated) deterioration of muscle and pulmonary function will also be evaluated. Any signs and symptoms experienced by the patient from the time of signing the informed consent through the final study visit will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter A. van Doorn, Prof. dr., Principal Investigator — Erasmus Medical Center; Nadine A.M.E. van der Beek, Dr., Principal Investigator — Erasmus Medical Center; Tim Preijers, Dr., Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared upon a reasonable request to the PI of the study.
Supporting Information: Study Protocol
Time Frame: These data will become available 3 months after the start of the trial.
Access Criteria: Upon a reasonable request